CLINICAL TRIAL: NCT05677633
Title: A Phase 1, Open-label Study to Validate Treatment-induced Biomarkers Following Sargramostim Treatment in Parkinson's Disease
Brief Title: Biomarker Validation Following Sargramostim Treatment in Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Partner Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0748-22-FB
Record Dates: First submitted 2022-12-15; First posted 2023-01-10 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Parkinson's Disease and Parkinsonism
Keywords: Leukine; sargramostim; biomarker
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leukine Treatment (Experimental): 48 week regimen of Leukine administered as a weight-based dose at 3 µg/kg/day for 5 days (week), followed by a 2-day holiday (weekend)
  Interventions: Drug: Sargramostim

INTERVENTIONS:
Drug: Sargramostim — Recombinant human GM-CSF produced by recombinant DNA technology using a yeast (S. cerevisiae) expression system
  Other Names: Leukine

SUMMARY:
Investigators will evaluate the safety of a 48 week regimen of Leukine administered as a weight-based dose at 3 ug/kg/ day for 5 days followed by a 2-day holiday. This 48 week long study will extend the prior biomarker evaluations observed in a previous study. Clinical signs and symptoms will be measured by personal well-being, physical, and neurological examinations (UPDRS Parts I, II, III, and IV assessments) and blood tests (CBC with differential, total T cell count, and a comprehensive metabolic sera panel). Leukapheresis will be performed to collect large numbers of immune cells for biomarker testing and immune phenotyping. Additionally, the investigators will determine whether immune deficits of PD are consistent during baseline data collection, and the potential Leukine-induced motor control and mobility improvements will be determined by UPDRS part I, II, III, and IV scores off treatment and on treatment.

DETAILED DESCRIPTION:
Primary Objectives:

There are two main study goals. First, the investigators will determine the safety of a 48 week regimen of Leukine administered as a weight-based dose at 3 µg/kg/day for 5 days, followed by a 2-day holiday. This 48 weeks (n=10) pilot study will continue to assess the safety of Leukine for treatment of Parkinson's disease (PD). Clinical signs and symptoms will be measured by personal well-being, physical, and neurological examinations (UPDRS Parts I, II, III, and IV assessments) and blood tests (CBC with differential, total T cell count, and a comprehensive metabolic sera panel). Due to fragility of the patient population and prior recorded adverse events the proposed dose reductions are justified. Second, in future preparations for an intended broader number of patient enrollments, the investigators wish to functionally examine any or all "putative" relevant biomarker assessments.

Secondary Objectives:

The investigators will examine over a time of 48 weeks, effects of treatment on defined adaptive immune deficits in PD as measured by analysis of peripheral blood mononuclear cells collected before and during Leukine therapy. The investigators will assess the individual T cell parameters that include links between T cell function and subset analyses and clinical neurological signs and symptoms. These immune parameters will be serially examined as they may contribute to the immune deficits in PD. Thus, timed analyses of changes in T cell phenotypes and/or function will be completed. In addition, the investigators will assess the functional stability of the immune deficits in PD. To this end, the investigators will examine T cell subsets in PD patients in this study against prior results. The investigators will determine whether the immune deficits of PD are consistent during baseline data collection. The investigators will evaluate the potential Leukine-induced motor control and mobility improvements by assessing UPDRS part I, II, III, and IV scores of treatment and on treatment. Additionally, over the course of this 48 week treatment study, investigators will also be assessing various biomarkers within plasma, peripheral blood, and the total lymphocyte and monocyte populations isolated from leukapheresis before Leukine therapy and after 24 and 48 weeks of treatment. Identified biomarkers will be correlated to disease severity and progression as assessed by UPDRS. Serum will also be collected to determine the generation of anti-drug neutralizing antibodies that may develop due to the dosing scheme.

ELIGIBILITY:
Inclusion Criteria:

1. Onset of bradykinesia and 1 or both of the following: rest tremor and/or rigidity
2. Asymmetric onset of clinical signs
3. Progressive motor symptoms
4. Age at onset 35-85 years
5. Duration of PD symptoms of at least 3 years
6. Female subjects must be either:

   1. Not pregnant, not breastfeeding, and not planning on becoming pregnant during the study;
   2. Not of childbearing potential, defined as one who has been postmenopausal for at least 1 year and with follicle stimulating hormone (FSH) levels in the laboratory defined postmenopausal range, or has been surgically sterilized, or has had a hysterectomy at least 3 months prior to the start of this trial; or
   3. If of childbearing potential, must agree to use an effective method of avoiding pregnancy to the end of the trial and must have a negative serum beta-human chorionic gonadotropin (β-HCG) test. Effective methods of avoiding pregnancy are contraceptive methods used consistently and correctly (including implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices, diaphragm with spermicide, male or female condoms with spermicide, or cervical cap), abstinence, or a sterile sexual partner.
7. Must be stage 4 or less according to the Hoehn and Yahr scale

Exclusion Criteria:

1. Atypical features indicative of a Parkinson-Plus disorder (Progressive Supranuclear Palsy (PSP), Multiple System Atrophy (MSA), Corticobasal Degeneration (CBD)) including cerebellar signs, supranuclear gaze palsy, apraxia and other cortical signs, or prominent autonomic failure
2. Neuroleptic treatment at time of onset of parkinsonism
3. Active treatment with a neuroleptic at time of study entry
4. History of repeated strokes with stepwise progression of parkinsonism
5. History of repeated head injury
6. History of definite encephalitis
7. More than one blood relative diagnosed with PD
8. Prominent gait imbalance early in the course (< 5 years)
9. Mini-mental state examination score <26
10. Hematological malignancy or coagulopathy
11. Abnormal blood analyses: hematocrit <30; white blood cell count >11.5; clinically significant laboratory data (e.g. alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 3x the upper limit of normal (ULN), or any abnormal laboratory value that could interfere with the assessment of safety in the judgment of the investigator; significant abnormalities on the clinical examination, vital signs, and clinical chemistry or hematology results (excluding findings of Parkinson's disease), that may interfere with the study or present a safety risk for the subject as judged by the clinical investigator charged in the care of study participants
12. Serious medical illness or co-morbidity that may interfere with participation in the study
13. Brain surgery for parkinsonism (DBS, cell implantation, gene therapy)
14. History of an autoimmune disorder or systemic inflammatory disorder deemed significant by physician
15. Immunostimulatory or immunosuppressive treatment (including amphetamines or systemic corticosteroids) within 90 days
16. Exclusively unilateral parkinsonism for longer than 3 years
17. Known hypersensitivity to granulocyte-macrophage colony-stimulating factor (GM-CSF), yeast-derived products
18. Current lithium treatment
19. Individuals with current diagnoses of alcohol or substance abuse/dependence
20. Anyone who is not appropriate for participation in this research protocol as deemed by the principal or co-investigator
21. Anyone who has previously been treated with granulocyte-macrophage colony-stimulating factor (GM-CSF) as an immunomodulatory therapy
22. Anyone with poor venous access
23. Anyone who has any illnesses or events that would cause a neurological abnormality, apart from Parkinson's disease.
24. Subjects with allergies or sensitivities to yeast products.
25. Subjects that have received a flu shot within the past 3 weeks.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Change in incidence of adverse events over time | every 6 months during the course of treatment, up to 48 weeks until drug cessation
  The safety of Leukine administration in PD will be examined by documenting abnormal results from complete blood count (CBC) with differential, total T cell count, or comprehensive metabolic panel analyses; abnormal physical and or neurological exam findings; abnormal levels of antibodies to Granulocyte-macrophage colony-stimulating factor (GM-CSF); clinically increasing Unified Parkinson's disease Rating Scale (UPDRS) part I, II, III, and IV scores as determined by the examining physician; and other adverse events. Adverse event logs will be reported every 4 weeks.

SECONDARY OUTCOMES:
Change in Treatment Biomarkers over time | every 6 months during the course of treatment, up to 48 weeks until drug cessation
  During the baseline visit and at 24 weeks and 48 weeks post-Leukine initiation, subjects will undergo leukapheresis to collect large amounts of monocytes and lymphocytes for biomarker evaluations. Cells will be harvested and subjected to proteomic and transcriptomic tests to assess therapeutic response and treatment-induced biomarkers. Biomarkers assessed will be proteins levels along with corresponding gene levels determined as fold change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Howard E Gendelman, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data with other researchers.

REFERENCES:
- [Background] Olson KE, Namminga KL, Lu Y, Schwab AD, Thurston MJ, Abdelmoaty MM, Kumar V, Wojtkiewicz M, Obaro H, Santamaria P, Mosley RL, Gendelman HE. Safety, tolerability, and immune-biomarker profiling for year-long sargramostim treatment of Parkinson's disease. EBioMedicine. 2021 May;67:103380. doi: 10.1016/j.ebiom.2021.103380. Epub 2021 May 14. PMID 34000620
- [Background] Abdelmoaty MM, Machhi J, Yeapuri P, Shahjin F, Kumar V, Olson KE, Mosley RL, Gendelman HE. Monocyte biomarkers define sargramostim treatment outcomes for Parkinson's disease. Clin Transl Med. 2022 Jul;12(7):e958. doi: 10.1002/ctm2.958. PMID 35802825
- [Background] Gendelman HE, Zhang Y, Santamaria P, Olson KE, Schutt CR, Bhatti D, Shetty BLD, Lu Y, Estes KA, Standaert DG, Heinrichs-Graham E, Larson L, Meza JL, Follett M, Forsberg E, Siuzdak G, Wilson TW, Peterson C, Mosley RL. Evaluation of the safety and immunomodulatory effects of sargramostim in a randomized, double-blind phase 1 clinical Parkinson's disease trial. NPJ Parkinsons Dis. 2017 Mar 23;3:10. doi: 10.1038/s41531-017-0013-5. eCollection 2017. PMID 28649610

DOCUMENTS (1):
  • Informed Consent Form (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT05677633/ICF_000.pdf